CLINICAL TRIAL: NCT04564027
Title: A Modular Phase 2a Multicentre Open-Label Study to Investigate DNA-damage Response Agents (or Combinations) in Patients With Advanced Cancer Whose Tumours Contain Molecular Alterations (PLANETTE)
Brief Title: A Study Investigating DNA-damage Response Agents in Molecularly Altered Advanced Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5339C00001; 2024-515102-12-00 (Registry Identifier: CTIS); 2020-002529-27 (EudraCT Number)
Record Dates: First submitted 2020-09-08; First posted 2020-09-25 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumours
Keywords: Ataxia telangiectasia mutated; Metastatic castration-resistant prostate cancer; Rad3-related protein
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — ceralasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Eligible participants (ATM altered AST), will receive oral dose of Ceralasertib as monotherapy.
  Interventions: Drug: Ceralasertib
- Cohort B (Experimental): Eligible participants (ATM altered mCRPC), will receive oral dose of Ceralasertib as monotherapy.
  Interventions: Drug: Ceralasertib

INTERVENTIONS:
Drug: Ceralasertib — Tablets will be administered orally
  Other Names: AZD6738

SUMMARY:
The study is investigating efficacy, safety and tolerability of DNA-damage Response Agents (or Combinations), in participants with advanced/metastatic solid malignancies whose tumours contain molecular alterations

DETAILED DESCRIPTION:
Current module of the study will consist of 2 cohorts as follows:

Cohort A (Advanced Solid Tumours [AST]): A total of ~25 molecularly eligible and centrally confirmed participants dosed at ceralasertib 160 mg twice daily will be enrolled into this cohort.

Cohort B (Metastatic castration-resistant prostate cancer [mCRPC]): A total of ~27 molecularly eligible and centrally confirmed participants dosed at ceralasertib 160 mg twice daily will be enrolled into Cohort B. Unfavourable circulating tumour cells (CTC) count requirement may be introduced for all participants to ensure an adequate (approximately ≥ 50%) number of participants with CTC count ≥ 5/7.5 mL blood.

The screening will have 2 parts, Part 1 and Part 2, which apply for both Cohort A and Cohort B.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a histologically confirmed diagnosis of AST (excluding NSCLC) or mCRPC tumour.
* Participants must have a deleterious or suspected deleterious ATM mutation in tumour or blood (germline or ctDNA). Definitions of qualifying ATM mutations may include deleterious/suspected deleterious, pathogenic/likely pathogenic, disease- or cancer-associated variants, or equivalent wording. Variants of unknown significance, benign or likely benign alterations are not qualifying.
* Participant must have normal organ and bone marrow function measured within 28 days prior to the first dose of study intervention.
* Participants who have no curative treatment options and are deemed appropriate for an investigational study in the opinion of the investigator.
* Availability of archival or fresh tumour specimens for central testing of ATM protein loss using immunohistochemistry and for confirmation of ATM mutation using next generation sequencing.
* Previously received and progressed on at least one novel hormonal agent (eg, abiraterone acetate, apalutamide, and/or enzalutamide) for the treatment of prostate cancer
* Participants with histologically confirmed metastatic castrate resistant prostate cancer.
* Documented prostate cancer progression at study entry while on androgen deprivation or after bilateral orchiectomy as assessed by the investigator.
* Serum testosterone levels ≤ 50 ng/dL (≤ 1.75 nmol/L) within (≤) 28 days before enrolment.

Exclusion Criteria:

* Any of the following cardiac diseases currently or within the last 6 months:

  1. Unstable angina pectoris.
  2. Congestive heart failure > Class 2 as defined by the New York Heart Association
  3. Acute myocardial infarction.
  4. Significant ventricular or supraventricular arrhythmias.
  5. Mean resting corrected QT interval (QTc) > 470 msec obtained from three electrocardiograms (ECGs) in 24 hours using the Fredericia formula.
  6. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, immediate family history of long QT syndrome or unexplained sudden death under 40 years of age.
  7. For Cohort B (mCRPC]), surgery or local prostatic intervention (excluding a prostatic biopsy) within 28 days of Cycle 1 Day 1.
* Participants with known active infections ((i.e., hepatitis B or C, tuberculosis, or COVID-19).
* Participants considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
* Participants with symptomatic and/or uncontrolled brain metastases.
* Previous therapy with an telangiectasia and rad3 related protein inhibitor.
* Exposure to a small molecule investigational product within 14 days or 5 half-lives.
* Concomitant use of known strong CYP 3A inhibitors and inducers.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (12):
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Tampa, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Ephrata, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Myrtle Beach, South Carolina
- France (4):
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Vandœuvre-lès-Nancy
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the requests portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5339C00001&attachmentIdentifier=4791fe13-fa2e-463d-89b8-f13b4123dbfa&fileName=247947_d5339c00001-csp_Final_Draft_to_approval_Redacted_16Apr24.pdf&versionIdentifier=
- See also: CSR Synopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5339C00001&attachmentIdentifier=c5913caa-a430-4d9b-a1d3-d55c7733c1c7&fileName=247947_CSR_synopsis_Final_Draft_to_approval__Redacted_16Apr24.pdf&versionIdentifier=
- See also: SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5339C00001&attachmentIdentifier=b13bf46a-762a-4d9a-a118-6f0b993cae41&fileName=247947_d5339c00001-SAP_Final_Draft_to_approval_Redacted_22Apr24_Final_format.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study from 01 December 2020 to 04 April 2023 at 18 centers in 3 countries.
Pre-assignment Details: The screening comprised of 2 parts, Part1 and Part 2, which applied for both Cohort A and Cohort B. Participants meeting the inclusion criteria were enrolled in the study. All the assessments were performed as per the schedule of the assessments.
Groups:
- Cohort A (aST): 240 mg of Ceralasertib: Participants with Ataxia telangiectasia mutated (ATM) altered Advanced solid tumour (aST) received 240 mg of ceralasertib twice daily from Day 1 to Day 14 of 28 days cycle.
- Cohort A (aST): 160 mg of Ceralasertib: Participants with ATM-altered aST received 160 mg of ceralasertib twice daily from Day 1 to Day 14 of 28 days cycle.
- Cohort B (mCRPC): 240 mg of Ceralasertib: Participants with ATM-altered Metastatic castration-resistant prostate cancer (mCRPC) received 240 mg of ceralasertib twice daily from Day 1 to Day 14 of 28 days cycle.
- Cohort B (mCRPC): 160 mg of Ceralasertib: Participants with ATM-altered mCRPC received 160 mg of ceralasertib twice daily from Day 1 to Day 14 of 28 days cycle.
Period: Overall Study
Arm/Group | Cohort A (aST): 240 mg of Ceralasertib | Cohort A (aST): 160 mg of Ceralasertib | Cohort B (mCRPC): 240 mg of Ceralasertib | Cohort B (mCRPC): 160 mg of Ceralasertib
Started | 8 | 30 | 1 | 15
Completed | 8 | 27 | 1 | 15
Not Completed | 0 | 3 | 0 | 0
Not completed — Ongoing treatment at Data cut off | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set consists of all participants who received at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (aST): 240 mg of Ceralasertib | Cohort A (aST): 160 mg of Ceralasertib | Cohort B (mCRPC): 240 mg of Ceralasertib | Cohort B (mCRPC): 160 mg of Ceralasertib | Total
Number analyzed (Participants) | 8 | 30 | 1 | 15 | 54
Age, Customized [Number; unit: Participants]
  18-64 years | 3 | 11 | 0 | 3 | 17
  65-84 years | 5 | 19 | 1 | 12 | 37
  ≥ 85 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 0 | 0 | 19
  Male | 3 | 16 | 1 | 15 | 35
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 0 | 0 | 0 | 0 | 0
  Native Hawaiin or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 8 | 11 | 0 | 6 | 25
  Not Reported | 0 | 7 | 0 | 4 | 11
  Missing | 0 | 9 | 0 | 5 | 14
  Other | 0 | 3 | 1 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 1 | 4
  Not Hispanic or Latino | 8 | 13 | 1 | 9 | 31
  Missing | 0 | 14 | 0 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Cohort A (aST): Objective Response Rate (ORR).
Description: ORR is defined as the percentage of participants who have at least one response of complete response (CR) or partial response (PR) prior to any evidence of progression (as defined by response evaluation criteria in solid tumours [RECIST] 1.1) that is confirmed at least 4 weeks later. The CR is defined as disappearance of all target and non-target lesions and no new lesions. The PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline and no new non-target lesion.
  Due to an increased frequency and early onset of Grade≥3 hematological toxicity noted among the participants receiving 240 mg of Ceralsertib, the sponsor decreased the dose to 160mg. Therefore, patients with the 240 mg BID starting dose were not included in the efficacy analyses for both study cohorts.
Time Frame: 2 years 4 months
Population: Evaluable for response set included all participants who were Molecularly Eligible Centrally Confirmed evaluable for response set with measurable disease at baseline and who received at least 1 dose of study intervention.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A (aST): 160 mg of Ceralasertib
Number analyzed (Participants) | 28
Percentage of participants | 7.14 [1.9 to 17.9]

2. Primary Outcome: Cohort B (mCRPC): Composite Response Rate.
Description: Composite response rate is defined as the investigator assessed radiological response by RECIST 1.1 for soft tissue and visceral lesions and Prostate Cancer Working Group 3 (PCWG3) for bone lesions, confirmed prostate specific antigen (PSA) decline of more than 50%, and/or confirmed circulating tumour cell [CTC] conversion from unfavorable (>=5 cells/7.5 ml blood) to favorable (<5 cells).
  Due to an increased frequency and early onset of Grade≥3 hematological toxicity noted among the participants receiving 240 mg of Ceralsertib, the sponsor decreased the dose to 160mg. Therefore, patients with the 240 mg BID starting dose were not included in the efficacy analyses for both study cohorts.
Time Frame: Up to 2 years 4 months
Population: Evaluable for response set included all participants who were Molecularly Eligible Centrally Confirmed evaluable for response set with measurable disease at baseline or unfavorable CTC count and who received at least 1 dose of study intervention.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort B (mCRPC): 160 mg of Ceralasertib
Number analyzed (Participants) | 13
Percentage of participants | 7.7 [0.8 to 26.8]

3. Secondary Outcome: Cohort A (aST): Duration of Radiological Response (DoR)
Description: DoR is defined as the time from the date of first documented response (confirmed CR/PR) until date of documented progression or death in the absence of disease progression.
Time Frame: Up to 2 years 4 months
Population: Molecularly eligible centrally confirmed evaluable for response set included all participants who were Molecularly Eligible Centrally Confirmed with measurable baseline disease and who received at least 1 dose of study intervention. The number of responders who subsequently progressed or died was 0, therefore, efficacy analysis was not conducted for Duration of response (DoR).
Arm/Group | Cohort A (aST): 160 mg of Ceralasertib
Number analyzed (Participants) | 0

4. Secondary Outcome: Cohort A (aST): Progression Free Survival (PFS)
Description: PFS is defined as the time from start of study intervention until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdraws from therapy or receives another anti-cancer therapy prior to progression. Progression is defined using (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  Due to an increased frequency and early onset of Grade≥3 hematological toxicity noted among the participants receiving 240 mg of Ceralsertib, the sponsor decreased the dose to 160mg. Therefore, patients with the 240 mg BID starting dose were not included in the efficacy analyses for both study cohorts.
Time Frame: Up to 2 years 4 months
Population: Molecularly eligible centrally confirmed set included all participants who were Molecularly Eligible Centrally Confirmed and who received at least 1 dose of study intervention.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Cohort A (aST): 160 mg of Ceralasertib
Number analyzed (Participants) | 28
Months | 3.7 [1.9 to 5.6]

5. Secondary Outcome: Cohort A (aST): Percentage Change in Tumor Size
Description: Percentage change in tumour size is defined as the reduction from baseline or the increase from baseline in the absence of a reduction in the sum of the longest diameters (or the short axis measurements for lymph nodes) of the target lesions. A negative change denotes a reduction in target lesion size.
Time Frame: Scan Visits 1 (Week 8), 2 (Week 16), 3 (Week 24), 4 (Week 32), 5 (Week 40), 6 (Week (48), 7 (Week 56)
Population: Molecularly eligible centrally confirmed evaluable for response set included all participants who were Molecularly Eligible Centrally Confirmed with measurable baseline disease and who received at least 1 dose of study intervention. Percentage change in tumor size was conducted every 8 weeks after the start of the treatment up to 1 year, then every 12 weeks until objective disease progression as per RECIST 1.1 or PCWG3 criteria.
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- Cohort A (aST): 240 mg of Ceralasertib: Participants with ATM -altered aST received 240mg of ceralasertib from Day 1 to Day 14 of 28 days cycle.
Arm/Group | Cohort A (aST): 160 mg of Ceralasertib | Cohort A (aST): 240 mg of Ceralasertib
Number analyzed (Participants) | 28 | 5
Percentage change
  Scan Visit 1 (Week 8): number analyzed (Participants) | 23 | 4
  Scan Visit 1 (Week 8) | 6.6 (22.45) | 6.2 (10.99)
  Scan Visit 2 (Week 16): number analyzed (Participants) | 13 | 1
  Scan Visit 2 (Week 16) | -4.7 (16.83) | 5.4 (NA) — Since there is only 1 participant with target lesion, descriptive statistics like Standard deviation cannot be calculated.
  Scan Visit 3 (Week 24): number analyzed (Participants) | 10 | 0
  Scan Visit 3 (Week 24) | -12.8 (21.47) |
  Scan Visit 4 (Week 32): number analyzed (Participants) | 5 | 0
  Scan Visit 4 (Week 32) | -17.9 (34.41) |
  Scan Visit 5 (Week 40): number analyzed (Participants) | 1 | 0
  Scan Visit 5 (Week 40) | -1.1 (NA) — Since there is only 1 participant with target lesion, descriptive statistics like Standard deviation cannot be calculated. |
  Scan Visit 6 (Week 48): number analyzed (Participants) | 1 | 0
  Scan Visit 6 (Week 48) | -100 (NA) — Since there is only 1 participant with target lesion, descriptive statistics like Standard deviation cannot be calculated. |
  Scan Visit 7 (Week 56): number analyzed (Participants) | 1 | 0
  Scan Visit 7 (Week 56) | -100 (NA) — Since there is only 1 participant with target lesion, descriptive statistics like Standard deviation cannot be calculated. |

6. Secondary Outcome: Cohort B (mRCPC): Percentage Change in Tumor Size
Description: Percentage change in tumour size is defined as the reduction from baseline or the increase from baseline in the absence of a reduction in the sum of the longest diameters (or the short axis measurements for lymph nodes) of the target lesions. A negative change denotes a reduction in target lesion size.
  Due to an increased frequency and early onset of Grade≥3 hematological toxicity noted among the participants receiving 240 mg of Ceralsertib, the sponsor decreased the dose to 160mg. Therefore, patients with the 240 mg BID starting dose were not included in the efficacy analyses for both study cohorts.
Time Frame: Scan Visits 1 (Week 8), 2 (Week 16), 3 (Week 24), 4 (Week 32)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Cohort B (mCRPC): 160 mg of Ceralasertib
Number analyzed (Participants) | 11
Percentage change
  Scan Visit 1 (Week 8): number analyzed (Participants) | 8
  Scan Visit 1 (Week 8) | 2.0 (21.35)
  Scan Visit 2 (Week 16): number analyzed (Participants) | 4
  Scan Visit 2 (Week 16) | -6.0 (9.37)
  Scan Visit 3 (Week 24): number analyzed (Participants) | 2
  Scan Visit 3 (Week 24) | -1.4 (11.75)
  Scan Visit 4 (Week 32): number analyzed (Participants) | 2
  Scan Visit 4 (Week 32) | -5.2 (13.21)

7. Secondary Outcome: Cohort A (aST) and B (mCRPC): Number of Participants With Serious and Non-serious Adverse Events
Description: The adverse events as a variable of safety and tolerability after admiration of ceralasertib was determined.
Time Frame: From Screening (Day -28 to Day -1) Until Follow-up (30 days post last dose), up to 2 years 4 months
Population: The safety analysis consists of all the participants who received at least 1 dose of ceralasterib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (aST): 240 mg of Ceralasertib | Cohort A (aST): 160 mg of Ceralasertib | Cohort B (mCRPC): 240 mg of Ceralasertib | Cohort B (mCRPC): 160 mg of Ceralasertib
Number analyzed (Participants) | 8 | 30 | 1 | 15
Participants
  All Adverse events (AE) | 8 | 30 | 1 | 15
  Any AE possibly related to treatment | 8 | 21 | 1 | 13
  Any AE of CTCAE Grade 3 or higher | 6 | 15 | 1 | 8
  Any AE of CTCAE Grade 3 or higher, possibly related to IP | 4 | 6 | 1 | 5
  Any AE with outcome of death | 0 | 0 | 1 | 0
  Any AE with outcome = death, possibly related to IP | 0 | 0 | 1 | 0
  Any SAE (including events with outcome = death) | 6 | 4 | 1 | 4
  Any SAE (including events with outcome = death), possibly related to IP | 3 | 2 | 1 | 1
  Any SAE leading to discontinuation of IP | 0 | 1 | 1 | 0
  Any SAE leading to discontinuation of IP, possibly related to IP | 0 | 0 | 1 | 0
  Any AE leading to discontinuation of IP | 0 | 1 | 1 | 1
  Any AE leading to discontinuation of IP, possibly related to IP | 0 | 0 | 1 | 1
  Any AE leading to dose modification | 4 | 10 | 1 | 5
  Any AE leading to dose reduction | 1 | 4 | 0 | 3
  Any AE leading to dose interruption | 4 | 7 | 1 | 3
  Any AE leading to dosing cycle delays | 1 | 0 | 0 | 1
  Any other significant AEs | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Screening (Day -28 to Day -1) Until Follow-up (30 days post last dose), up to 2 years 4 months
Description: Safety analysis consist of all participants who received at least 1 dose of study intervention.
Arm/Group | Cohort A (aST): 240 mg of Ceralasertib | Cohort A (aST): 160 mg of Ceralasertib | Cohort B (mCRPC): 240 mg of Ceralasertib | Cohort B (mCRPC): 160 mg of Ceralasertib
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/30 | 1/1 | 0/15
Serious Adverse Events (participants affected / at risk) | 6/8 | 4/30 | 1/1 | 4/15
Other Adverse Events (participants affected / at risk) | 8/8 | 30/30 | 1/1 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (aST): 240 mg of Ceralasertib (N=8) | Cohort A (aST): 160 mg of Ceralasertib (N=30) | Cohort B (mCRPC): 240 mg of Ceralasertib (N=1) | Cohort B (mCRPC): 160 mg of Ceralasertib (N=15)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (aST): 240 mg of Ceralasertib (N=8) | Cohort A (aST): 160 mg of Ceralasertib (N=30) | Cohort B (mCRPC): 240 mg of Ceralasertib (N=1) | Cohort B (mCRPC): 160 mg of Ceralasertib (N=15)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 6 (8) | 8 (10) | 0 (0) | 6 (8)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 6 (8) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | 1 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 4 (8) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Dysguesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scleral haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5) | 1 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 9 (9) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 7 (7) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (9) | 1 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 13 (14) | 0 (0) | 8 (10)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (6) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 3 (5) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 4 (7) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 2 (4) | 1 (1) | 1 (1)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 7 (7) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 8 (8) | 1 (2) | 5 (5)
oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mucosal discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anorectal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB. Access to this document must be restricted to relevant parties.

DOCUMENTS (2):
  • Study Protocol (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT04564027/Prot_005.pdf
  • Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT04564027/SAP_001.pdf